CLINICAL TRIAL: NCT03922373
Title: The Single-dose and Multiple-dose Pharmacokinetic Study of Benzonatate Soft Capsule in Chinese Healthy Subjects
Brief Title: A Study of Benzonatate Soft Capsule in Chinese Healthy Subjects
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: CSPC ZhongQi Pharmaceutical Technology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EY20170502
Record Dates: First submitted 2018-10-31; First posted 2019-04-19 (Actual); Last update posted 2019-04-19 (Actual); Status verified 2019-04

CONDITIONS: Cough
MeSH Terms: conditions — Cough

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Benzonatate (Experimental)
  Interventions: Drug: Group A: Benzonatate 100mg; Drug: Group B: Benzonatate 200mg; Drug: Group C: Benzonatate 400mg

INTERVENTIONS:
Drug: Group A: Benzonatate 100mg — Subjects in group A will be given benzonatate 100mg once after a 10-hour fast in the first day of the trail
Drug: Group B: Benzonatate 200mg — Subjects in group B will be given benzonatate 200mg once after a 10-hour fast in the first day of the trail, and they will be given benzonatate 200mg thrice in the second and third day of the trail, in the fourth day, they will be given benzonatate 200mg once after a 10-hour fast.
Drug: Group C: Benzonatate 400mg — Subjects in group C will be given benzonatate 400mg once after a 10-hour fast in the first day of the trail

SUMMARY:
Objective to study the pharmacokinetic, safety and efficacy of Single-dose and multiple-dose of benzonatate in Chinese healthy male and female subjects.

DETAILED DESCRIPTION:
Objective to study the pharmacokinetic, safety and efficacy of Single-dose and multiple-dose of benzonatate in Chinese healthy male and female subjects. The study was designed to be single-center, open, and parallel, there are 3 groups A, B, C, each group will be enrolled in 12 healthy adult subjects. Single-dose of pharmacokinetics will be carried out in group A and C, single-dose and multiple-dose of pharmacokinetics will be carried out in group B. Subjects in group A and C will be given benzonatate of 100mg and 400mg respectively, Subjects in group B will be given benzonatate of 200mg. Subjects in group A and C will be given benzonatate once after a 10-hour fast in the first day of the trail. Subjects in group B will be given benzonatate once after a 10-hour fast in the first day of the trail, and they will be given benzonatate thrice in the second and third day of the trail, in the fourth day, they will be given benzonatate once after a 10-hour fast. After completing blood collection and safety inspection at the appropriate time points, subjects can leave the test center. The main pharmacokinetic parameters will be calculated, to fully reflect the characteristics of drug absorption, distribution, metabolism and excretion in human body. The main pharmacokinetic parameters include Tmax, Cmax, Css, AUC0-t, AUC0-∞, λz, t1/2, Vd/F, CL/F, and so on.

ELIGIBILITY:
Inclusion Criteria:

* 1. You should fully understand the testing content, process and adverse reaction. Freely given informed consent.

  2. Male or Female ages 18 through 45 (include 18 and 45).

  3. The male subjects weighed more than 50 kg, the female subjects weighed more than 45kg. Body Mass Index(BMI) between 18 and 28, BMI=Weight(kg)/Height2(m2).

Exclusion Criteria:

* 1. Allergy to benzonatate, allergic constitution (Allergic to a variety of medicines and foods).

  2. Abnormal physical examination and abnormal vital signs, and have clinical significance.

  3. Abnormal results of laboratory studies and have clinical significance. 4. Abnormal electrocardiogram and have clinical significance. 5. The hepatitis B surface antigen(HbsAg), hepatitis C antibody, HIV antibody and antigen, Treponema pallidum antibody（TP-Ab）were positive.

  6. Patients with cardiovascular system, urinary system, digestive system, nervous system, respiratory system, mental or immunodeficiency diseases.

  7. Dysphagia or with gastrointestinal history influencing drug absorption. 8. Patients with any diseases that increase the risk of bleeding (e.g. acute gastritis, duodenal ulcer, and so on).

  9. Patients smoked more than 5 cigarettes a day in the first 3 months of screening 10. Alcohol breath test were positive (blood-alcohol concentration>0.0mg/100ml) , or have history of alcoholism (more than 14 units of alcohol every week, 1 unit is equal to 285ml of beer, 25ml of spririts, or 100ml of wine.

  11. Drug abuse screening were positive by urinalysis, or have a history of substance abuse or taken drugs last 3 years.

  12. Subjects (or his fere) have family planning in the next 3 months, or can't take effective contraceptive measures in the next 3 months.

  13. Female subjects during lactation, the quantitative of β-HCG exceed the upper limit of normal range.

  14. Donate blood or massive blood loss (>450ml) in the first 3 months of screening.

  15. Taken any drugs that can inhibit the activity of liver enzyme in the first 28 days of screening, or taken the inhibitor or inducer of CYP3A4, P-gp, Bcrp, such as Itraconazole, Ketoconazole, Dronedarone.

  16. Taken any prescription drugs, OTC, vitamin products or Chinese herbal medicine in the first 14 days of screening.

  17. Special diets (e.g. pitaya, mango, pomelo) or strenuous exercise in the first 14 days of screening, or other factors to influence drug absorption, distribution, metabolism and excretion.

  18. Have attended clinical trial in the first 3 months of screening 19. The patient can't finish the study according to protocol requirements. 20. Acute disease or simultaneous medication between screening stage and the first time taking study drugs.

  21. Have consumed any alcoholic or caffeinated food or beverage such as chocolate and coffee in the first 48 hours of taking the study drug.

  22. Investigator believes other factors not suitable for testing.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2018-09-10 (Actual); Primary Completion 2019-02-27 (Actual); Study Completion 2019-04-30 (Estimated)

PRIMARY OUTCOMES:
Tmax | day 1 and day 4
  Time to peak
Cmax | day 1 and day 4
  peak plasma concentration
t1/2 | day 1 and day 4
  elimination half-life time
AUC0-t | day 1 and day 4
  Area under the plasma concentration versus time curve from the medication to the last time the concentration can be measured
AUC0-∞ | day 1 and day 4
  Area under the plasma concentration versus time curve from the medication extrapolate the infinity time
CL/F | day 1 and day 4
  elimination ratio

CONTACTS AND LOCATIONS:
Overall Officials: Yang Lin, M.D., Principal Investigator — Beijing Anzhen Hospital; Shan Jing, M.D., Principal Investigator — Beijing Anzhen Hospital
Locations (1):
- Cspc Nbp Pharmaceutical.Co.Ltd, Shijiazhuang, Hebei, China

IPD SHARING:
Plan to Share IPD: Yes